CLINICAL TRIAL: NCT01097811
Title: Erythromycin Versus Neomycin Treatment for Overt Hepatic Encephalopathy: a Double-blind, Randomised, Controlled Trial.
Brief Title: Comparison Between Erythromycin and Neomycin Treatment of Hepatic Encephalopathy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: UPECLIN HC FM Botucatu Unesp (Other)
Collaborators: Biophisics Department of Biosciences Institute - Unesp (Unknown); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Fernando Gomes Romeiro / Doctor, Faculdade de Medicina de Botucatu - UNESP
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: upeclin/HC/FMB-Unesp-41
Record Dates: First submitted 2010-03-31; First posted 2010-04-02 (Estimated); Last update posted 2010-04-28 (Estimated); Status verified 2010-04

CONDITIONS: Hepatic Encephalopathy; Hypertension, Portal; Liver Cirrhosis
Keywords: Hepatic Encephalopathy; Hypertension, Portal; Liver Cirrhosis; Bacterial Overgrowth Syndrome
MeSH Terms: conditions — Hepatic Encephalopathy; Hypertension, Portal; Liver Cirrhosis; Blind Loop Syndrome | interventions — Erythromycin; Neomycin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Erythromycin (Active Comparator)
  Interventions: Drug: Erythromycin
- Neomycin (Active Comparator)
  Interventions: Drug: Neomycin

INTERVENTIONS:
Drug: Erythromycin — 250 mg orally q.i.d.
  Arms: Erythromycin
Drug: Neomycin — 1 g orally q.i.d.
  Arms: Neomycin

SUMMARY:
Comparison between the efficacy of two different antibiotics in patients with overt hepatic encephalopathy. The study is randomized, controlled and double-blinded.

ELIGIBILITY:
Inclusion Criteria:

* Hepatic cirrhosis or portal hypertension
* Hepatic Encephalopathy

Exclusion Criteria:

* Acute liver failure
* Neuropsychiatric diseases
* Inflammatory bowel diseases
* Intestinal obstruction
* Shock
* Renal insufficiency
* Alcoholic hepatitis
* Alcohol abuse
* Antibiotic premedication

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2008-06; Primary Completion 2010-06 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Recovery of hepatic encephalopathy | three years
  comparison of efficacy between two drugs for the treatment of hepatic encephalopathy

SECONDARY OUTCOMES:
length of hospitalization caused by hepatic encephalopathy | three years
  comparison of efficacy between two drugs for reducing the length of hospitalization during treatment of hepatic encephalopathy

CONTACTS AND LOCATIONS:
Overall Officials: Fernando G Romeiro, Principal Investigator — Faculdade de Medicina de Botucatu, Unesp; Carlos A Caramori, Study Chair — Faculdade de Medicina de Botucatu, Unesp
Locations (1):
- Faculdade de Medicina de Botucatu - Universidade Estadual Paulista, Botucatu, São Paulo, Brazil